CLINICAL TRIAL: NCT04059653
Title: Primary Care Evaluation of A Novel Disposable Neuromuscular Electrical Stimulation Treatment For Female Urinary Incontinence: A Randomised Controlled Trial
Brief Title: Evaluation of a New Technology for the Treatment of Bladder Leakage in Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID19 pandemic. Cannot recruit from primary care during pandemic
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Jackie Oldham, Professor Jackie Oldham, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R123366; 223014 (Other: IRAS)
Record Dates: First submitted 2019-08-07; First posted 2019-08-16 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Urinary Incontinence; Urinary Incontinence, Stress; Urinary Incontinence, Urge
Keywords: neuromuscular electrical stimulation; incontinence
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress; Urinary Incontinence, Urge | interventions — Electric Stimulation; Therapeutics

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Electrical stimulation (Experimental): Neuromuscular electrical stimulation treatment
  Interventions: Device: Electrical stimulation
- Treatment As Usual (Active Comparator): Usual GP treatment
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Device: Electrical stimulation — Electrical stimulation device
  Arms: Electrical stimulation
Other: Treatment as usual — GP treatment as usual
  Arms: Treatment As Usual

SUMMARY:
Evaluation of a new technology for the treatment of bladder leakage in women. The objective is to compare quality of life and other incontinence associated outcomes between women receiving routine General Practitioner (GP) prescribed care for urinary incontinence compared with those prescribed the electrical stimulation device.

DETAILED DESCRIPTION:
This United Kingdom study will comprise a single blind, primary care, post-market evaluation of a novel neuromuscular electrical stimulation treatment for urinary incontinence . Women with GP determined urinary incontinence (urgency, stress or mixed) will be randomised into one of two groups (intervention or control). The control group will receive routine care via their GP practice. The intervention group will receive the electrical stimulation device. Treatment will last for 12 weeks with a Quality of Life (QoL) primary end point immediately post treatment with a second phase to explore the impact of a further 12 weeks maintenance programme in the intervention group compared to routine care. There will be a further two year follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Aged between 18 and 65
* GP determined urinary incontinence

Exclusion Criteria:

* Abnormal abdominal mass
* Clinical history of urinary retention problems
* Severe atrophic vaginitis, vaginal infection, vaginal lesion, severe urogenital prolapse at the level of the vaginal introitus or any other pathology of the vagina or labia
* Pregnancy or given birth within the last three months
* Implanted pacemaker
* Recent pelvic surgery (within the last 12 months)
* Recent haemorrhage, haematoma and/or tissue damage to the vagina
* Undergoing any active therapy or review appointments for pelvic malignancy
* Current urinary tract infection confirmed by urinary dip stick test on initial visit (can be included following a subsequent clear urinary dipstick test)
* Manual dexterity insufficient to place the electrical stimulation device in the vagina
* Presence of a severe neurological conditions such as Multiple Sclerosis, Motor Neuron Disease or Parkinson's Disease
* Multiple co-morbidities to the extent that the activities involved in the pad test (i.e. stair climbing) cannot be completed
* Insufficient cognitive ability to provide informed consent and/or participate in the study
* Unwillingness to participate in the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Condition specific quality of life | 12 weeks
  The primary outcome measure is Quality of Life measured through self-completion of the short form version of the International Consultation on Incontinence Questionnaire-Urinary Incontinence (ICIQ-UI). The Short Form is a brief and psychometrically robust patient-completed questionnaire for evaluating the frequency, severity, and impact on urinary incontinence in research and clinical practice across the world.
  Scoring & analysis: Question items include: frequency of urinary incontinence, amount of leakage and leak interference. The overall score is calculated from the sum of:
  Leak frequency (minimum 0, maximum 5) Leak amount (minimum 0, maximum 6) Leak interference (minimum 0, maximum 10) Overall score is therefore between 0-21 - the higher the score the worse the outcome

SECONDARY OUTCOMES:
Female Sexual Function Index (FSFI) | 12 weeks
  Brief questionnaire measure of sexual functioning in women. It was developed for the specific purpose of assessing domains of sexual functioning (e.g. sexual arousal, orgasm, satisfaction, pain) in clinical trials.
  The individual domain scores and full scale (overall) score of the FSFI are derived by adding the scores of the individual items that comprise each domain and multiplying the sum by a domain factor. The six domain scores are added together to obtain the full-scale score. Within the individual domains, a domain score of zero indicates that the subject reported having no sexual activity during the past month.
  Desire: Minimum score 1 maximum 5 Arousal: Minimum score 0 maximum 5 Lubrication: Minimum score 0 maximum 5 Orgasm: Minimum score 0 maximum 5 Satisfaction: Minimum score 0 maximum 5 Pain: Minimum score 0 maximum 5
  Score are multiplied by pre defined factors with a total range of between 2 and 36 where 36 is the most satisfied
Sexual dysfunction questionnaire | 12 weeks
  The International Urogynecological Association Pelvic Organ Prolapse / Urinary Incontinence Sexual Questionnaire to assess sexual function.
  To score the sub-scales of which there are six in sexually active women and four in women who are not sexually active, half of the items must be answered, imputation is not recommended, and either mean calculation or transformed sum methods are recommended. There is a detailed process for calculating total scores that runs to three pages that has been published and validated in the International Urogynaecology Journal 2013
Patient Global Impression of Severity and of Improvement | 12 weeks
  A well-validated global assessment of improvement questionnaire for women with urinary stress incontinence
  Scoring and analysis: The severity part of the scale is a single question asking the patient to rate how their urinary tract condition is now on a scale of 1 = Normal to 4 = Severe. The improvement part of the scale is a single question asking the patient to rate how their urinary tract condition is now compared with how it was before they started the study on a scale of 1 = very much better to 7 = very much worse
1-hour in-clinic provocative pad weight test | 12 weeks
  A standardised Food and Drug Administration recommended test
  A standardised one hour test protocol is adopted from the recommendations of the International Continence Society.
  Scoring and analysis: Volume of urine leaked over one hour calculated from the difference in pad weight pre and post 1-hour activities.
  In terms of reporting the severity of urine loss is considered cured (<2g / hour), mild (2-10g / hour), moderate (11-50g/hour) and severe >50g/hour).
User experience Diaries | 12 weeks
  A diary that records user experience will be completed every two weeks over the 12 weeks of the study.
  A second diary that records usability specific to treatment arm will be completed every other day in the first four weeks of the study and then every week for the following eight weeks.

OTHER OUTCOMES:
Health economics | 12 weeks
  Although a formal Health Economic analysis is not part of the protocol, data to enable such an analysis will be collected. Participants will be asked to complete a diary of expenditure on incontinence products during the week preceding each assessment point.

CONTACTS AND LOCATIONS:
Overall Officials: Jackie Oldham, PhD, Principal Investigator — Univeristy of Manchester; Sheila McCorkindale, MBChB FRCGP, Study Chair — University of Manchester
Locations (1):
- South Manchester GP Federation, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oldham J, Herbert J, McBride K. Evaluation of a new disposable "tampon like" electrostimulation technology (Pelviva(R)) for the treatment of urinary incontinence in women: a 12-week single blind randomized controlled trial. Neurourol Urodyn. 2013 Jun;32(5):460-6. doi: 10.1002/nau.22326. Epub 2012 Sep 28. PMID 23023996
- See also: Improving quality of life for women. Providing groundbreaking technology for the treatment of urinary incontinence — https://www.femeda.com